CLINICAL TRIAL: NCT03075111
Title: Field Study of Host-based Immunoassay for Differentiating Bacterial From Viral Infections (Post-marketing Study of ImmunoXpert™ - SPIRIT Study)
Brief Title: Host-based Immunoassay for Differentiating Bacterial From Viral Infections (Post-marketing Study of ImmunoXpert™ - SPIRIT Study)
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MM-1007-SP
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ImmunoXpert — Host based immune response test distinguishing viral versus bacterial infection

SUMMARY:
This is a retrospective external field study of a novel in vitro diagnostic (IVD) assay (ImmunoXpert™).

The study will involve reviewing the medical charts of about 4500 pediatric patients that were tested using ImmunoXpert™ as part of the routine workup for acute febrile illness.

ImmunoXpert™ uses a computer algorithm to combine immunoassay measurements of three host immune proteins (TRAIL, IP-10, and CRP) present in human blood. The test is intended for use in conjunction with clinical assessments and other laboratory findings as an aid to differentiate bacterial from viral infection.

Statistical analysis will be performed to compare the diagnostic accuracy of ImmunoXpert™ with that of current practice lab testing e.g., WBC, CRP, and PCT (whichever were taken as part of routine care) and clinical suspicion at time of requisition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 month to 18 years that were admitted due to acute febrile illness, and ImmunoDx test was taken as part of their workup.

The febrile illness should also fulfill the following criteria:

* The patient had a peak temperature ≥38°C (AND)
* Symptoms initiated ≤ 7 days before sampling (AND)
* A retrospective diagnosis of bacterial or viral or mixed infection was anonymously determined by a panel of three independent senior pediatricians.

The non-infectious disease control group will include:

* A retrospective diagnosis of a non-infectious disease was anonymously determined by a panel of three independent senior pediatricians physicians.
* Patients with a non-infectious disease ( and ImmunoDx test was wrongly taken)

Exclusion Criteria:

* Samples from patients who had one or more of the following criteria will be excluded from the study:
* Another infection episode during the last 3 weeks before sampling
* Congenital immune deficiency (CID)
* A proven or suspected HIV-1, HBV, HCV infection
* Active hematological malignancy
* Current treatment with immune-suppressive or immune-modulating therapies including without limitations:
* Use of high dose steroids >1 mg/kg/day prednisone or equivalent in the last two weeks
* Monoclonal antibody administration
* Intravenous immunoglobulin (IVIG)
* Other illnesses that affect life expectancy and/or quality of life
* Suspicion of gastrointestinal infection

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Patients with an acute bacterial infection
  2. Patients with an acute viral infection
  3. Patients with an acute co-infection (bacterial and viral)
  4. Patients with an undetermined disease etiology
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2015-11-07 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of a host-response based diagnostics in differentiating between bacterial and viral etiology of patients with an acute febrile disease. | 0-7 days after the initiation of symptoms

SECONDARY OUTCOMES:
The sensitivity and specificity of a host-response based diagnostics in differentiating between infectious and non-infectious disease etiology | 0-7 days after the initiation of symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hillel Yaffe Medical center, Hadera
  - Bnei Zion medical center, Haifa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein A, Shapira M, Lipman-Arens S, Bamberger E, Srugo I, Chistyakov I, Stein M. Diagnostic Accuracy of a Real-Time Host-Protein Test for Infection. Pediatrics. 2023 Dec 1;152(6):e2022060441. doi: 10.1542/peds.2022-060441. PMID 37916266